CLINICAL TRIAL: NCT01033656
Title: An Open, Randomized Study Treating Refractory Adult-onset Still's Disease With Interleukin-1 Receptor Antagonist Anakinra (Kineret), Compared to an Established, Single Anti-rheumatic Drug Treatment
Brief Title: Treatment of Refractory Adult-onset Still's Disease With Anakinra: a Randomized Study
Acronym: NordicAOSD05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Uppsala University Hospital (Other); Helse Stavanger HF (Other Government); Tampere University Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Kuopio University Hospital (Other); Jyväskylä Central Hospital (Other); Satakunta Central Hospital (Other); University Hospital, Umeå (Other); University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Dan Nordstrom, ass.prof, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NordicAOSD05; 2005-003173-24 (Other: EudraCT)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Adult-Onset Still's Disease
Keywords: adult-onset Still's disease; anakinra; prednisolone; disease-modifying antirheumatic drug; methotrexate; efficacy; patients
MeSH Terms: conditions — Still's Disease, Adult-Onset | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; Methotrexate; Azathioprine; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): experimental drug of study
  Interventions: Drug: anakinra
- comparator (Active Comparator): comparators:methotrexate, azathioprine, leflunomide or supfasalazine
  Interventions: Drug: comparators

INTERVENTIONS:
Drug: anakinra — 100 mg subcutaneous injection daily
  Other Names: Interleukin-1 receptor antagonist
  Arms: Anakinra
Drug: comparators — po drugs, comparators
  Other Names: methotrexate, azathioprine, leflunomide, sufalalazine
  Arms: comparator

SUMMARY:
An open, randomized, parallel-group, comparative, multicentre study. Patients on corticosteroids (plus conventional therapy) will be randomized to receive anakinra (Kineret®), or one of the following: methotrexate, azathioprine, leflunomide, cyclosporin A or sulphasalazine. Patients enter the study if considered refractory to corticosteroids (prednisolone equivalent ≥10 mg/day) at the time of randomization.

The randomized phase of the study will be followed by an open-label extension (OLE) phase, to follow-up drug survival, efficacy, tolerability and disease-related parameters of long-term treatment with anakinra or one of the study DMARDs or a combination of study drugs for additional 28 weeks.

DETAILED DESCRIPTION:
Product: Kineret (anakinra) Comparative agents: Methotrexate or azathioprine or leflunomide or cyclosporin A or sulphasalazine Protocol title: An open, randomized study treating refractory adult-onset Still's disease with IL-1ra anakinra (Kineret, compared to an established, single anti-rheumatic treatment Target Disease: Adult-onset Still's disease Patients: 23 patients diagnosed with AOSD, living in the four Nordic countries.

Study Objectives: To follow the changes in clinical status and disease activity in patients receiving anakinra, compared to those treated with an established DMARD, in addition to corticosteroids in patients with refractory AOSD. To compare the changes in disease-related parameters (global health, patient's assessment on disease, laboratory values) in the two randomized groups. To assess the safety of anakinra in AOSD. To follow-up drug survival, efficacy, tolerability and disease-related parameters of long-term treatment in AOSD (open phase).

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with AOSD according to preliminary classification by Yamaguchi (1992).
* Other diseases with similar symptoms must be excluded. Has been exposed to a corticosteroid for ≥2 months prior to randomization for AOSD.
* Needs a prednisolone dose ≥10 mg/day or equivalent, yet unacceptable disease activity determined by the investigator.
* Anti-TNF agents must be discontinued 4 to 8 weeks prior to commencing study medication.

Exclusion Criteria:

* Use of corticosteroids (prednisolone equivalent <10 mg/day.
* History of recurrent or chronic infection, including:

  * tuberculosis
  * any malignancy
  * any other major chronic inflammatory disease syndrome
  * drug or alcohol abuse
  * known positivity for hepatitis B, C or HIV.
* Use of anti-TNF agents during ≤4 weeks (etanercept) or≤8 weeks (infliximab or adalimumab) prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of patients reaching remission of the disease, after eight weeks of the randomized study treatment (Remission: afebrile and normalization of acute phase reactants) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan C Nordstrom, MD, PhD, Principal Investigator — Helsinki University Hospital, Department of Medicine
Locations (1):
- Ann Kataja Knight, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordstrom D, Knight A, Luukkainen R, van Vollenhoven R, Rantalaiho V, Kajalainen A, Brun JG, Proven A, Ljung L, Kautiainen H, Pettersson T. Beneficial effect of interleukin 1 inhibition with anakinra in adult-onset Still's disease. An open, randomized, multicenter study. J Rheumatol. 2012 Oct;39(10):2008-11. doi: 10.3899/jrheum.111549. Epub 2012 Aug 1. PMID 22859346